CLINICAL TRIAL: NCT06301178
Title: Effect of Vitamin D Injection on Hypertrophic Scars and Keloids
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12548
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Dermatologic Disease
MeSH Terms: conditions — Skin Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D deficiency (Active Comparator): patients with vitamin D deficiency or insufficiency (<12 ng/ml and 12-19 ng/ml, respectively) received systemic and intralesional vitamin D injections
  Interventions: Drug: Cholecalciferol
- vitamin D sufficiency (Active Comparator): Patients with vitamin D sufficiency (20 and greater ng/mL) of vitamin D received only intralesional injections of vitamin D on hypertrophic scars and keloids.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Vitamin D has various critical regulatory roles, including inflammatory control, cellular proliferation and differentiation, and wound healing regulation.

SUMMARY:
Scars and keloids cause patients severe morbidity and psychological distress. Hypertrophic scars rise above the skin but stay within the scar boundaries, while keloids expand.

The development of keloids and hypertrophic scars is a consequence of insufficient wound healing. These lesions are distinguished by excessive ECM deposition. Excessive ECM deposition is caused by increased inflammatory and proliferative processes and decreased remodeling activities. These scarring lesions are also linked to genetic and systemic causes

ELIGIBILITY:
Inclusion Criteria:

- Age from 12 years to 50 years. Patients with hypertrophic scars and keloids

Exclusion Criteria:

Age below 12 years and above 50 years. Patients received other treatment modalities for hypertrophic scars and keloids.

Systemic and other skin diseases. Patients were already receiving supplemental vitamin D.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Clinical scoring by Vancouver Scale Score | 3 months
  Four characteristics of the scar are assessed. These are: vascularity, height, pliability, and pigmentation. Each characteristic is given a score, which are added together to give an overall score between 0 and 13

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine-Fayoum university, Al Fayyum, Egypt

REFERENCES:
- [Derived] Hassan AR, Binsaleh AY, El-Tahlawi SM, El-Amir AM, Ishak MM, Alsubaie N, El-Masry TA, Bahaa MM, Eldesoqui M, Kamal M. Impact of Vitamin D Injection on Keloids and Hypertrophic Scars. J Cosmet Dermatol. 2025 Apr;24(4):e70118. doi: 10.1111/jocd.70118. PMID 40135774